CLINICAL TRIAL: NCT00915408
Title: A Phase I Dose Escalation Study of the Combination of Lenalidomide (Revlimid®), Dexamethasone and Cyclophosphamide in Patients Refractory or Relapsing From Stable Disease With Multiple Myeloma
Brief Title: A Dose Escalation Study of the Combination of Lenalidomide (Revlimid®), Dexamethasone and Cyclophosphamide in Patients Refractory or Relapsing From Stable Disease With Multiple Myeloma
Acronym: CRD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Dr Steve Schey, King's College Hospital NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05CC15; REC - 06/Q1606/75; EudraCT - 2005-005145-19
Record Dates: First submitted 2009-06-05; First posted 2009-06-08 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2013-04

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Cyclophosphamide; Dexamethasone; Lenalidomide
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; Dexamethasone; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CRD (Experimental)
  Interventions: Drug: Lenalidomide; Drug: Dexamethasone; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Lenalidomide — Oral lenalidomide 25mg daily on Days 1-21 every 28 days cycles for up to 9 cycles. From Cycle 10 Lenalidomide 25mg orally on days 1-21, every 28 days.
  Other Names: Revlimid
Drug: Dexamethasone — Dexamethasone 20mgs orally, daily on Days 1-4 and 8-11 repeated every 28 day cycles for up to 9 cycles.
Drug: Cyclophosphamide — Oral Cyclophosphamide will be added to the regime starting on days 1 and 8. The dose of Cyclophosphamide will be escalated in cohorts rising in 100mg increments from 300 to 700mgs days 1,and 8 every 28 day cycles for up to 9 cycles.

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose (MTD) and to evaluate the safety of cyclophosphamide when given on days 1 and 8 in a 28 day cycle in doses starting at 300mg ranging to 700mg in combination with Lenalidomide (Revlimid®) plus dexamethasone in patients who present with relapsed or refractory myeloma.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign an informed consent form.
2. Age >18 years at the time of signing the informed consent form.
3. Proven diagnosis of multiple myeloma.
4. Relapse or Refractory disease with evidence of progression after at least 2 cycles of anti-myeloma treatment.
5. Relapse or refractory disease with evidence of progressive disease after at least 1 previous therapy this may include consolidation of induction with a stem cell transplant).
6. Subjects may have been previously treated with thalidomide and/or radiation therapy. In addition, radiation therapy initiated prior to or at baseline (Day 1) must be complete prior to the initiation of therapy. The initiation of radiation therapy after baseline (Day 1) will be considered to be a treatment failure (except when given to treat or to promote the healing of a pathological fracture).
7. Measurable levels of myeloma paraprotein in serum (>5 gms/L) or urine > 2 g excreted in a 24-hour collection sample).
8. Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1 or 2.
9. Able to adhere to the study visit schedule and other protocol requirements.
10. Women of childbearing potential (WCBP) must have a negative serum or urine pregnancy test within 10 - 14 days and again within 24 hours of starting study drug. In addition, sexually active WCBP must agree continued abstinence from heterosexual intercourse or to use adequate contraceptive methods starting 4 weeks prior to the initiation of therapy. WCBP must agree to have pregnancy tests weekly for the first 4 weeks, then monthly while on study drug (every 14 days for women with irregular cycles) and 4 weeks after the last dose of study drug. Men must also agree to use a condom if their partner is of child bearing potential, even if they have had a successful vasectomy.
11. Disease free of prior malignancies for equal to or over 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in-situ" of the cervix or breast.
12. Able to receive low dose aspirin (e.g. 75mg) as prophylactic anticoagulant medication to prevent thromboembolism unless contraindicated. If low dose aspirin is contraindicated, subjects will receive another form of anticoagulant prophylaxis according to hospital guidelines.

Exclusion Criteria:

1. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
2. Pregnant or lactating females.
3. Any of the following laboratory abnormalities:

   1. Absolute neutrophil count (ANC) <1.000 cells/mm3 (1.0 x 109/L)
   2. Platelet count <.75.000/mm3 (75 x 109L)
   3. Serum creatinine >2.5 mg/dL (221 umol/L)
   4. Serum SGOT/AST or SGPT/ALT >3.0 x upper limit of normal (ULN)
   5. Serum total bilirubin >2.0 mg/dL (34 umol/L)
4. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
5. Known hypersensitivity to thalidomide, dexamethasone or cyclophosphamide.
6. Prior history of uncontrollable side effects to dexamethasone therapy
7. The development of a desquamating rash while taking thalidomide
8. Any prior use of Lenalidomide (Revlimid®)
9. Use of any standard/experimental anti-myeloma drug therapy within 28 days of entry or use of any experimental non-drug therapy (e.g. donor leukocyte/mononuclear cell infusions) within 56 days of entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2006-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity defined as: a) NCI Grade 4 haematological toxicity b) NCI Grade ¾ non-haematological toxicity | Weekly for first cycle
Safety (type, frequency, severity, and relationship of adverse events) | Weekly for first cycle then monthly

SECONDARY OUTCOMES:
Time to progression | Monthly
Paraprotein response | Monthly
Bone marrow response | Baseline, end of treatment and disease progression
Duration of response | Monthly
Overall survival | Monthly

CONTACTS AND LOCATIONS:
Overall Officials: Steve Schey, FRCP FRACP FRCPath, Principal Investigator — King's College Hospital NHS Trust
Locations (2):
- United Kingdom (2):
  - King's College Hospital NHS Foundation Trust, London
  - Royal Marsden NHS Foundation Trust, London